CLINICAL TRIAL: NCT02617394
Title: Comparing Two Ultrasound-based Methods to Assess Diaphragm Movement
Brief Title: Novel vs. Traditional US Diaphragm Scanning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00060267
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Diaphragm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Diaphragm scanning - traditional method first
- Study group (Experimental)
  Interventions: Other: Diaphragm scanning - novel method first

INTERVENTIONS:
Other: Diaphragm scanning - traditional method first — The first (pre-block) diaphragm scan with ultrasound will be done on both sides using the liver (right side) and spleen (left side) as acoustic windows. The second (post-block) diaphragm scan will be done on both sides using a novel method in which lung sliding is used as a guide to identify the diaphragm and quantify diaphragm thickening upon respiration.
  Arms: Control group
Other: Diaphragm scanning - novel method first — The first (pre-block) diaphragm scan with ultrasound will be done on both sides using a novel method in which lung sliding is used as a guide to identify the diaphragm and quantify diaphragm thickening upon respiration. The second (post-block) diaphragm scan will be done will be done on both sides using the liver (right side) and spleen (left side) as acoustic windows.
  Arms: Study group

SUMMARY:
Occasionally, doctors need to be able to see whether the diaphragm - a muscle in the chest that helps control breathing - is moving properly. If the diaphragm is paralyzed or not moving properly, this can affect a person's breathing. After certain nerve blocks - where a part of the body is frozen using local anesthetic - the nerve controlling diaphragm movement can be anesthetized, causing diaphragm paralysis. Ultrasound can be used to see the diaphragm and measure its movement, but the easiest and fastest way to do this is debatable. The investigators wish to compare two ultrasound-based methods to image diaphragm movement to see which one offers the quickest and easiest way to determine if the diaphragm is paralyzed.

DETAILED DESCRIPTION:
Background and rationale The diaphragm muscle helps to control breathing: upon inhalation, the diaphragm contracts, helping to draw air into the lungs. Air is exhaled when the diaphragm relaxes. Measurement of diaphragmatic movement is an important tool in assessing function of the diaphragm. With the introduction of ultrasound technology to the bedside, the motion of the diaphragm and lungs can be visualized in real time. This affords practitioners the ability to detect when the diaphragm is paralyzed or is not moving properly. For example, the phrenic nerve, which controls diaphragm movement, is often anesthetized during interscalene brachial plexus block. As a result, the diaphragm on the block side is paralyzed, compromising breathing. This can have serious implications for patients who already suffer from respiratory difficulties.

There are several previously described methods for assessing diaphragm movement using ultrasound. The investigators wish to compare two methods to determine which one is more user-friendly and offers the fastest time to measure diaphragm movement. The first method will rely on the ability to identify and image the right and left diaphragms through the acoustic windows of the liver and spleen, respectively, and then record diaphragm movement in M-mode. The second method will rely on the ability to identify the location of the diaphragm by imaging lung sliding, followed by re-orientation of the ultrasound probe to enable measurement of changes in diaphragm thickness with respirations. The investigators hypothesize that, due to the more obvious visibility of the structures involved, the second method will result in more accurate confirmation of diaphragm paralysis.

Study objectives The primary objective is to determine which of two ultrasound-based methods of imaging the diaphragm offers the fastest and easiest way to confirm diaphragm paralysis. A secondary objective is to determine the inter-rater reliability among two individuals using the same scanning method.

Hypothesis The investigators hypothesize that imaging lung sliding with ultrasound followed by diaphragm thickness measurement will be easier and faster for practitioners to detect diaphragm motion/paralysis.

Study procedures Following informed written consent, eligible patients will be recruited in the University of Alberta pre-admission clinic (PAC) or day ward. Once the patient arrives in the block area, a study investigator will scan the patient's diaphragm on both sides using one of the two scanning methods. The scanning method to be used will be determined randomly; the investigator will be given a sealed envelope containing brief instructions on the method of diaphragm imaging to be used. The investigator will scan one side of the patient and then the other side. The order of scanning will be left to the participating investigator. A study team member will record the length of time taken for the investigator to obtain what they deem to be optimal images, which will be saved on the ultrasound machine. Following this, the regional block will be administered.

Once the regional block is deemed to be working, the second set of diaphragm scans will be done. A study investigator will be given brief instructions on how to perform the scanning method, which will be the same one done pre-block. Again, time taken to obtain optimal images will be recorded, and the images will be saved on the ultrasound machine. This will end the study procedure, and the patient will be transferred to the operating theater.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years of age or older)
* Provided informed consent
* Supraclavicular block indicated for surgical anesthesia

Exclusion Criteria:

• Refusal to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Time taken to image diaphragm | Approximately 2-5 minutes from start of ultrasound scan
  Total time will be from when the probe is placed on the patient's body to when a good quality image of the diaphragm is recorded. This will be done on each side of the body.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Houston JG, Morris AD, Howie CA, Reid JL, McMillan N. Technical report: quantitative assessment of diaphragmatic movement--a reproducible method using ultrasound. Clin Radiol. 1992 Dec;46(6):405-7. doi: 10.1016/s0009-9260(05)80688-9. No abstract available. PMID 1493655
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830